CLINICAL TRIAL: NCT04398459
Title: A Phase II, Multicenter, Open-label Trial to Determine the Safety and Efficacy of Ibrutinib in Refractory/Relapsed Autoimmune Hemolytic
Brief Title: The Safety and Efficacy of Ibrutinib in Refractory/Relapsed Autoimmune Hemolytic Anemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Jun Shi, Director, Regenerative Medicine Clinic Center, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020005
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Refractory/Relapsed Autoimmune Hemolytic Anemia
Keywords: Ibrutinib; BTK Inhibitor; autoimmune hemolytic anemia; AIHA
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iBRIAN (Experimental)
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Each recruited subject will accept Ibrutinib treatment.
  Other Names: BTK inhibitor

SUMMARY:
This is an open-label, single-arm study to evaluate the safety and efficacy of Ibrutinib in subjects with refractory/relapsed autoimmune hemolytic anemia.

ELIGIBILITY:
Inclusion Criteria:

* ECOG ≤ 3
* Age from 6 to 70.
* Diagnosed with WAIHA or MAIHA.
* Meets the criteria of relapsed / refractory AIHA.
* Meets the criteria of DAT-negative AIHA without any other inherited or acquired hemolytic diseases, and previously treated effectively with glucocorticoids and rituximab.
* Signed informed consent.
* Organs in good function.

Exclusion Criteria:

* Nursing woman
* Active bacterial, virus, fungal or parasitic infection, including HIV infection, HbsAg and HBV DNA positive, HCV DNA positive, etc.
* Diagnosed with cold agglutinin disease or cold agglutinin syndrome or paroxysmal cold hemoglobinuria.
* Secondary AIHA caused by drugs or infection.
* Received rituximab in 8 weeks before enrollment.
* Previously received treatment with BTK inhibitor.
* Previously received organ or stem cell transplantation.
* Have a history of thrombosis or organ infarction.
* Diagnosed with an active stage of connective tissue disease.
* Have a history of lymphoproliferative tumors or any other malignant tumors.
* Have other inherited or acquired hemolytic diseases.
* Received low-molecular-weight heparin or warfarin within 1 week before enrollment or during the Ibrutinib treatment.
* Received CYP3A4 Enzyme Inhibitors or Inducers within 1 week before enrollment or during the Ibrutinib treatment.
* Have a history of mental illness.
* Inability to understand or to follow study procedures.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | within 12 weeks

SECONDARY OUTCOMES:
Incidence of adverse events and severe adverse events | within 48 weeks
Relapse free survival rate | within 48 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Zhoukou Central Hospital, Zhoukou, Henan
  - The Second Affilated Hospital of Shandong First Medical University, Tai’an, Shandong
  - Regenerative Medicine Center, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fang LW, Pan H, Shi J. [Ibrutinib treatment for 2 cases of relapsed/refractory autoimmune hemolytic anemia: a pilot study]. Zhonghua Xue Ye Xue Za Zhi. 2020 May 14;41(5):412-416. doi: 10.3760/cma.j.issn.0253-2727.2020.05.009. Chinese. PMID 32536139